CLINICAL TRIAL: NCT06702475
Title: Are There Sleep-related Factors That Contribute to an Increased Incidence of Pre-eclampsia
Brief Title: Are There Sleep-related Factors That Contribute to an Increased Incidence of Pre-eclampsia at Altitude?
Status: Not yet recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, David Patz, Senior Clinical Instructior, Pulmonary Medicine., University of Colorado, Denver
Other Study IDs: 23-1743
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Pre-Eclampsia
Keywords: Pre-Eclampsia, Altitude, Sleep Apnea
MeSH Terms: conditions — Pre-Eclampsia; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pregnant with pre-eclampsia at altitude (Cohort 1): Pregnant women at High Country Obstetric Clinic in Summit County Colorado (about 9000 ft.) who develop pre-eclampsia.
  Home sleep testing with Watch PAT-one will be done soon after diagnosis of pre-eclampsia.
  Up to 20 in this cohort
  Interventions: Diagnostic Test: Home Sleep Test with Watch PAT-one
- healthy pregnant women at altitude (Cohort 2): Pregnant healthy women at High Country Obstetric Clinc in Summit County Colorado will also be studied with the Watch PAT-one home sleep test..
  Up to 20 will be chosen to match the subjects, 1 by 1, in cohort 1, regarding gestational time of the home sleep test, and match age, pre-pregnant BMI, and race as best as available of the volunteered subjects. Up to another 20 pregnant healthy women at altitude may be recruited, not matching a subject in cohort 1, to have Watch PAT-one home sleep testing in the 33rd to 34th week of pregnancy.
  Interventions: Diagnostic Test: Home Sleep Test with Watch PAT-one
- healthy pregnant women at sea level (Cohort 3): Up to 40 healthy pregnant women at sea level, in vicinity of Baltimore, will be recruited to have Watch PAT-one home sleep testing, matching the subjects in cohort 2 regarding gestational time of testing, Race, Age and pre-pregnant BMI as best as available.
  Interventions: Diagnostic Test: Home Sleep Test with Watch PAT-one

INTERVENTIONS:
Diagnostic Test: Home Sleep Test with Watch PAT-one — Each participant will have a Watch-PAT one home sleep test, recording pulse oximetry, pulse tonometry, wrist actigraphy, snoring (by microphone), and chest motion by accelerometer.

SUMMARY:
Women at altitude have an increased incidence of pre-eclampsia. Populations at altitude have a greater incidence of sleep apnea. And women with sleep apnea are at increased risk of developing preeclampsia. This research project will recruit for home sleep testing: healthy pregnant women at altitude (Summit County , Colorado at 9000 ft.), and women with preeclampsia at altitude, in order to learn whether either sleep apnea or nocturnal hypoxemia is more common or more severe in women with preeclampsia, than in healthy women at altitude. In addition a healthy co-hort of pregnant women will be studied at sea level, to compare to the healthy cohort of pregnant woman in Summit County, to learn to degree that this difference in altitude effects the severity of sleep apnea and hypoxemia.

DETAILED DESCRIPTION:
It is known that high altitude increases the risk of preeclampsia and small for gestational age births. Our questions are: 1). Is sleep apnea during pregnancy more common and/or more severe at altitude? And 2) Do the women who develop preeclampsia at altitude have more severe sleep apnea, or worse hypoxemia during sleep, than the women at altitude who do not develop preeclampsia. We will perform WatchPAT-one home sleep tests (PAT = peripheral arterial tonometry) on up to 20 pregnant women in Summit County Colorado (>9000 ft.elevation) who develop preeclampsia during pregnancy (soon after diagnosis), and also on up to 20 pregnant healthy women in Summit County, and 20 healthy pregnant women in Baltimore (at sea level). These healthy pregnant women in Summit County and Baltimore will be selected from volunteer participants, to best match age, pre-pregnancy BMI, and race with individuals in Summit County who are studied with preeclampsia and they will be studied at the gestational timing that matches their Summit County preeclampsia matching subject. In addition to the up to 20 healthy pregnant subjects at Summit County and 20 in Baltimore, who match the preeclampsia subjects, we will recruit up to 20 more in Summit County and 20 more in Baltimore, to study specifically in the 33rd or 34th gestational week, to improve our ability to evaluate the effects of altitude on sleep apnea, during pregnancy. Information on the births, including height and weight and apgar scores will be assessed, in part to see whether sleep apnea during pregnancy affects outcomes. All sleep studies will be scored at the JHH (Johns Hopkins Hospital) Bayview sleep lab's Center for Interdisciplinary Sleep Research and Education.

ELIGIBILITY:
Inclusion Criteria: pregnant, age 18-35, possession of, or availablitiy of using a cell phone.

-

Exclusion Criteria: for the control group the following are exclusion criteria: hypertension, known sleep apnea, asthma requiring daily inhaler use, other lung disease, diabetes

For the group who are recruited at the time of diagnosis of pre-eclampsia - hypertension is not an exclusion criteria.

-

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women, age 15-35, some who are healthy, and some who have developed preeclampsia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea index 4% | in a single full night recording
  number of apneas and hypopneas dropping oxygen saturation 4%, per hour

OTHER OUTCOMES:
Apnea-Hypopnea Index 3% | in a single full night recording
  number of apneas and hypopneas dropping oxygen saturation 3%, per hour
Central Apnea-Hypopnea Index 4% | in a single full night recording
  number of central apnea or hypopnea events dropping oxygen saturation 4%, per hour
Central Apnea Hypopnea Index 3% | in a single full night recording
  number of centrap apnea or hypopnea events dropping oxygen saturation 3%, per hour
Mean Oxygen Saturation during sleep | averaged through one full night recording
  the average oxygen saturation
Lowest oxygen saturation during sleep | during one full night recording
  the single lowest oxygen saturation measured
Time (in minutes) with oxygen saturation below 89% | during one full night recording
  as above
Time (in minutes) with oxygen saturation below 85% | during one full night recording
  as above
percentage of babies small for gestational age | measurements made at birth. Correlations will be determined at completion of research study
  length weight and gestational age will be considered for each baby, to determine if it is small for gestational age. comparison will be made between cohorts. But also, analysis to determine is AHI correlated with "small for gestational age"
Apgar at 1 minute | Measurement, 1 minute after birth. Correlations will be determined at completion of research study.
  This will be looked at for correlation with the AHI, along with the usual comparison between cohorts
Apgar at 5 minutes | Measurement, 5 minutes after birth. Correlations will be determined at completion of research study
  This will be looked at for correlation with the AHI, along with the usual comparison between cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Argani, MD, Study Chair — Johns Hopkins Hospital OB-GYN

IPD SHARING:
Plan to Share IPD: Undecided
The data will likely be shared. The precise mechanism of sharing the data is not yet determined.